CLINICAL TRIAL: NCT03419468
Title: LCI-GER-NOS-TAB-001: Pilot Study of a Tablet to Administer the Cancer-Specific Geriatric Assessment (CSGA) in Geriatric Patients With Cancer
Brief Title: LCI-GER-NOS-TAB-001: Tablet for Geriatric Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LCI-GER-NOS-TAB-001; 00023842 (Other: Advarra IRB)
Record Dates: First submitted 2018-01-11; First posted 2018-02-05 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2021-02

CONDITIONS: Self Geriatric Assessment Measure (SGAM)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): iPad administration of Self Geriatric Assessment Measure (SGAM)
  Interventions: Other: Self Geriatric Assessment Measure (SGAM)
- 2 (Active Comparator): Paper survey administration of Self Geriatric Assessment Measure (SGAM)
  Interventions: Other: Self Geriatric Assessment Measure (SGAM)

INTERVENTIONS:
Other: Self Geriatric Assessment Measure (SGAM) — Self Geriatric Assessment Measure

SUMMARY:
The Self Geriatric Assessment Measure [SGAM] is based on a standard diagnostic tool used to evaluate geriatric cancer patients in order to determine the appropriateness of cancer directed therapy at LCI. This questionnaire has sections that matches portions of a self-administered geriatric assessment in patients aged 70 or older with malignancy. The prolonged duration of time needed to complete the assessment makes its performance less feasible in standard practice settings.

In previously published studies the Cancer Specific Geriatric Assessment (CSGA) has been provided both via written questionnaire and by personal computer in subjects 70 years of age or older. With improvements in technology, the goal is to evaluate the feasibility of administering the SGAM via an iPad tablet and compare results to both gold standard paper format and prior desktop computer data.

This study proposes the use of an iPad tablet to administer the SGAM may help:

Improve the completion rate of the SGAM assessment Reduction in the time of completion Improvement in the accuracy of reporting

DETAILED DESCRIPTION:
Primary Objective

Assess and compare the proportions of subjects completing, defined as recording responses for at least 70% of actionable questions of the Self Geriatric Assessment Measure (SGAM) in subjects aged 70 years or older with malignancy using an iPad tablet versus written questionnaire.

Secondary Objectives

To assess and compare the proportions of subjects completing the SGAM without assistance using an iPad tablet versus written questionnaire.

To evaluate and compare the total times of interaction with the SGAM using an iPad tablet versus written questionnaire in both all evaluable subjects and the subset of evaluable subjects completing the SGAM.

To evaluate and compare the distributions of percentages of recorded responses on actionable questions (from 0% to 100%) on the SGAM using an iPad tablet versus written questionnaire in both all evaluable subjects and the subset of evaluable subjects completing the SGAM.

To describe the rate of technical issues experienced by iPad survey users.

To assess and compare the completion rates and times to completion of the gold standard written format.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following criteria:

* At least 70 years of age
* Histologically or cytologically confirmed malignancy within the past 1 year
* Ability to read and understand English
* Willingness to complete either tablet or paper based assessment independently and without assistance from caregiver, if applicable
* Willingness and ability to understand and sign a written informed consent document

Exclusion Criteria

Subjects must not meet any of the following criteria:

* Any prior history of whole brain radiation therapy for known brain metastasis
* Known cerebrovascular event within the last 4 weeks from enrollment
* Known to be legally blind or has a history of severe hearing loss that could impair ability to complete questionnaire in the opinion of the investigator

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 89 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-18 (Actual)

PRIMARY OUTCOMES:
Survey completion rate | 12 months
  Assess and compare the proportions of subjects completing, defined as recording responses for at least 70% of actionable questions of the SGAM in subjects aged 70 years or older with malignancy using an iPad tablet versus written questionnaire.

SECONDARY OUTCOMES:
Rate of survey completion without assistance | 12 months
  To assess and compare the proportions of subjects completing the SGAM without assistance using an iPad tablet versus written questionnaire.
Total time of interaction with iPad survey | 12 months
  To evaluate and compare the total times of interaction with the SGAM using an iPad tablet versus written questionnaire in both all evaluable subjects and the subset of evaluable subjects completing the SGAM.
Percentage of recorded responses | 12 months
  To evaluate and compare the distributions of percentages of recorded responses on actionable questions (from 0% to 100%) on the SGAM using an iPad tablet versus written questionnaire in both all evaluable subjects and the subset of evaluable subjects completing the SGAM.
Rate of technical issues within iPad group | 12 months
  To describe the rate of technical issues experienced by iPad survey users.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Haggstrom, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT03419468/ICF_000.pdf